CLINICAL TRIAL: NCT05163015
Title: Impact of Oncogeriatric Consultation on Quality of Life of Patients Aged 75 and More With Cancer
Acronym: ONCOGERIA-QDV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-009-ONCOGERIA-QDV
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-01

CONDITIONS: Cancer
Keywords: Cancers; aged patients; oncogeriatric consultation; quality of life
MeSH Terms: conditions — Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with oncogeriatric consultation: with oncogeriatric consultation" group: patients aged 75 and more with cancer with oncogeriatric consultation
  Interventions: Other: Data collection
- without oncogeriatric consultation: without oncogeriatric consultation" group: patients aged 75 and more with cancer without oncogeriatric consultation
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Description: quality of life assessment

SUMMARY:
Among patients with cancer, 6 in 10 are over 65 years of age. In order to improve quality of life of aged cancer patients, the oncogeriatric consultation has been created. Oncogeriatric consultation aim to help oncologists determine the best solutions to combine therapy and quality of life. Factors influencing quality of life of cancer patients have been studied previously. However, these studies always focus on one specific cancer.

DETAILED DESCRIPTION:
The aim of the study is to study factors associated with quality of life in patients aged 75 and more with cancer, notably the oncogeriatric consultation.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged of 75 and more
* with cancer
* with indication of oncogeriatric consultation according G8
* agreeing to participate in the study

Exclusion Criteria:

-less than 75 years old

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged of 75 and more with cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 | Day 0
  The QLQ-C30 is a generic questionnaire with 30 questions coded in 4 response modalities (not at all (1), a little (2), enough (3), a lot (4)) or in 7 response modalities (from very bad (1) to excellent ( 7)).
  Questions are summarized in five multiitem domains (physical, role, cognitive, emotional, and social functioning) and nine single item domains (fatigue, pain, nausea/vomiting, appetite loss, financial impact; diarrhea, constipation, sleep disturbance and quality of life).
  Each domain is scored between 0 and 100. For functional domains, a high score value represents a high level of quality of life. For symptom domains, a high score represents an important level of symptoms (a low level of quality of life).
EORTC QLQ-C30 | Day 60
  The QLQ-C30 is a generic questionnaire with 30 questions coded in 4 response modalities (not at all (1), a little (2), enough (3), a lot (4)) or in 7 response modalities (from very bad (1) to excellent ( 7)).
  Questions are summarized in five multiitem domains (physical, role, cognitive, emotional, and social functioning) and nine single item domains (fatigue, pain, nausea/vomiting, appetite loss, financial impact; diarrhea, constipation, sleep disturbance and quality of life).
  Each domain is scored between 0 and 100. For functional domains, a high score value represents a high level of quality of life. For symptom domains, a high score represents an important level of symptoms (a low level of quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Godinot, Reims, Grand Est, France

IPD SHARING:
Plan to Share IPD: No